CLINICAL TRIAL: NCT05937009
Title: Effects of Orientation Exercise Program on Older Adults, Motor Skills, Cognitive and Emotional State: a Pilot Study
Brief Title: 12 Weeks Orienteering Program Exercise on Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Franclim Martins, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Franclim Martins
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-07

CONDITIONS: Community-dwelling Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental Orienteering group program (Experimental): The experimental group intervention will attend the orienteering program. The program integrates 3 sessions / week during 12 consecutive weeks.
  Interventions: Other: Orienteering exercise program
- The control group (No Intervention): The control group will maintain the usually daily activities, not attending any exercise program.
  After study end, the control group will have the opportunity to participate on an exercise program.

INTERVENTIONS:
Other: Orienteering exercise program — Orienteering exercise program running for 12 weeks (30-45 minutes, 3 sessions/week). Sessions will have 4 phases: 1) Signature of attendance sheet; 2) warm-up exercises for 5 minutes; 3) Start of orienteering proofs, where the departs will occur individually, with 3 interval minutes between participants; 4) stretches session, to return to a calm state.
  Arms: Experimental: Experimental Orienteering group program

SUMMARY:
This study aims to determine the effects of an orientation exercise program addressed to old on physical-motor, cognitive, and affective competencies.

This quasi-experimental study is a controlled trial involving an orientation exercise program. The program will run for 12 weeks (3 sessions per week).

Participants will be clustered into two groups: the experimental group will perform the exercise orientation sessions, and the control group will maintain regular activities routines. Evaluations will be performed before and after the intervention.

After the study is finished, the control group will attend a similar exercise program.

DETAILED DESCRIPTION:
The aging process is lived for all and is associated with uncountable limitations, such as physical, psychological, cognitive, or emotional, that daily translate into difficulty in accomplishing normal activities (2). Simple tasks such as getting up and sitting, carrying a shopping bag, or climbing some stairs, start being seen as an obstacle, much because of aging and the associated decline in physical and cognitive competencies such as balance, limb strength, aerobic capacity, motor coordination, processing speed, memory, executive functioning and, consequently, affective competences, such as emotional states and depression may also be compromised (1).

Despite the above, it is known that there are some ways and alternatives that, even not reversing the aging process, might delay it, promoting healthy aging (6). Scientific advances recommend regular physical exercise since exercise ensures a more active lifestyle and, therefore, a less dependent on others' life. There are many options that physical exercise professionals can choose for planning physical exercise programs for older people (3).

Nonetheless, instead of exercise planning training prescription, other options can be used to achieve healthy aging. In alternative to traditional exercise training, sporting modalities, such as orientation, may benefit this population.

According to a study, after applying a protocol that included changes to the terrain to improve older adults' balance, there were significant improvements in their stride time (4).

Other studies done within the same area, which applied one questionnaire on functional well-being, and four scales on depression, gastrointestinal system, physical activity, and healthy index to senior athletes between the ages of 67 and 71, found significant improvements in all the referred parameters except for the depression scale where the control group made up of older adults who do not practice the modality showed better results (5).

However, the literature is scarce concerning the participation in orientation programs by the elderly population, namely in terms of this program's effect on aerobic capacity, lower limb strength, motor coordination, processing speed, memory, and executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-75 years old;
* Locomotor independent capacity;
* Independent living in the community;
* Historical of physical activity practice;
* Attended, at least, the 3º school grade.

Exclusion Criteria:

* Cognitive impairment such < 15 points in Mini-Mental State Examination (MMSE);
* Evidence of neuromuscular disturb;
* Use of medication that conditions the performance of the orientation exercise tasks.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from the beginning, between groups comparison, in physical competencies | 0, 12 weeks
  Fullerton Advance Balance Scale to assess balance, ranging from 0 (worst) to 40 (best) points
Change from the beginning, between groups comparison, in physical competencies | 0, 12 weeks
  Senior Fitness Test, 6 minutes walking to assess aerobic capacity, measure in meters
Change from the beginning, between groups comparison, in physical competencies | 0, 12 weeks
  Senior Fitness Test, Sit and Stand to assess limb strength, measure by the number of repetitions
Change from the beginning, between groups comparison, in physical competencies | 0, 12 weeks
  Soda Pop Test to assess motor coordination.
Change from the beginning, between groups comparison, in cognitive competencies | 0, 12 weeks
  Trail Making Test (Part A and B) to assess processing speed and executive functioning, measure in seconds
Change from the beginning, between groups comparison, in cognitive competencies | 0, 12 weeks
  Rey Auditory Verbal Test to assess memory, measure in seconds
Change from the beginning, between groups comparison, in affective competencies | 0, 12 weeks
  Profile of Mood States to assess mood states, ranging from -32 (best) to 200 (worst) points
Change from the beginning, between groups comparison, in affective competencies | 0, 12 weeks
  Geriatric Depression Scale to assess depression state, ranging from 0 (best) to 30 (worst) points

SECONDARY OUTCOMES:
Cognitive impairment | 0 weeks
  Mini-Mental State Examination, ranging from 0 (worst) to 30 (best) points

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Pereira, Doctoral degree, Principal Investigator — University of Évora; José Marmeleira, Doctoral degree, Principal Investigator — University of Évora
Locations (1):
- Universidade de Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bliss ES, Wong RH, Howe PR, Mills DE. Benefits of exercise training on cerebrovascular and cognitive function in ageing. J Cereb Blood Flow Metab. 2021 Mar;41(3):447-470. doi: 10.1177/0271678X20957807. Epub 2020 Sep 20. PMID 32954902
- [Background] Eckstrom E, Neukam S, Kalin L, Wright J. Physical Activity and Healthy Aging. Clin Geriatr Med. 2020 Nov;36(4):671-683. doi: 10.1016/j.cger.2020.06.009. Epub 2020 Aug 19. PMID 33010902
- [Background] Hemmeter UM, Ngamsri T. [Physical Activity and Mental Health in the Elderly]. Praxis (Bern 1994). 2022;110(4):193-198. doi: 10.1024/1661-8157/a003853. German. PMID 35291872
- [Background] McCarthy, I., Suzuki, T., Tyler, N. & Holloway, C. (2016). Mobility in the built environment: Age-related changes in gait characteristics when walking on complex terrain. Healthy Aging Research, 5:10.
- [Background] Ostlund-Lagerstrom L, Blomberg K, Algilani S, Schoultz M, Kihlgren A, Brummer RJ, Schoultz I. Senior orienteering athletes as a model of healthy aging: a mixed-method approach. BMC Geriatr. 2015 Jul 8;15:76. doi: 10.1186/s12877-015-0072-6. PMID 26152308
- [Background] Thomas E, Battaglia G, Patti A, Brusa J, Leonardi V, Palma A, Bellafiore M. Physical activity programs for balance and fall prevention in elderly: A systematic review. Medicine (Baltimore). 2019 Jul;98(27):e16218. doi: 10.1097/MD.0000000000016218. PMID 31277132